CLINICAL TRIAL: NCT01251406
Title: A Randomized, Parallel, Placebo-controlled, Double-blind Phase IIa Study of Efficacy and Safety of Recombinant Human Neuregulin-1 (Neucardin) in Subjects With Stable Chronic Heart Failure
Brief Title: Efficacy and Safety of Human Neuregulin-1 to Treat Stable Chronic Heart Failure
Acronym: ZS-01-210
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Collaborators: Zensun USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-01-210
Record Dates: First submitted 2010-11-17; First posted 2010-12-01 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Chronic Heart Failure
Keywords: Stable; Chronic Heart Failure; Systolic
MeSH Terms: conditions — Systolic Murmurs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subcutaneous administration for daily for 8 hours a day for 10 days
  Interventions: Drug: Placebo
- rhNRG-1 Dose 1 (Experimental): Subcutaneous administration for daily for 8 hours a day for 10 days
  Interventions: Drug: rhNRG-1 Dose 1
- rhNRG-1 Dose 2 (Experimental): Subcutaneous administration for 8 hours a day for 10 days
  Interventions: Drug: rhNRG-1 Dose 2

INTERVENTIONS:
Drug: Placebo — Daily subcutaneous administration for 8 hours a day for 10 days
  Other Names: Placebo: 0 dose
  Arms: Placebo
Drug: rhNRG-1 Dose 1 — Daily subcutaneous administration for 8 hours a day for 10 days
  Other Names: Neucardin
  Arms: rhNRG-1 Dose 1
Drug: rhNRG-1 Dose 2 — Daily subcutaneous administration for 8 hours a day for 10 days
  Other Names: Neucardin
  Arms: rhNRG-1 Dose 2

SUMMARY:
The mortality of chronic heart failure patients remains high. Recombinant human Neuregulin-1 (rhNRG-1, also called Neucardin) is a 61 amino acid peptide that acts directly on damaged heart muscle cells to restore their structure and function. This study will investigate the safety and efficacy of rhNRG-1 to treat stable chronic heart failure.

DETAILED DESCRIPTION:
This randomized, parallel, placebo-controlled, double-blind, multi-center study will assess the safety and efficacy of rhNRG-1 also known as Neucardin as a treatment for stable chronic heart failure.

A total of 120 subjects, who have chronic heart failure with a NYHA classification of II or III, and are on a stable regimen of ACEI/angiotensin receptor blocker (ARB), beta-blocker, and/or diuretic for at least 3 months prior to receiving study medication and anticipated to remain on the stable regimen through the treatment period can enroll as per specific inclusion and exclusion criteria.

Subjects will be hospitalized for 10 days during the treatment period and will be infused subcutaneously with rhNRG-1 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Male or female subjects.
* Have chronic heart failure defined as NYHA classification of II or III.
* Be on a stable regimen of ACEI/ARB and/or beta-blocker 3 months prior to receiving study medication and are expected to remain on a stable HF medication regime throughout the duration of the trial.
* Left ventricular ejection fraction (LVEF) of < 35% as determined at screening by 2-D echocardiography.
* Is able to understand and provide informed consent.
* If subject has dilated cardiomyopathy, ischemic heart disease or corrected valvular heart disease, and had surgery to repair or replace value, the surgery must have been performed 3 months prior to receiving study medication and the surgical area is functioning normally.
* Proper birth control must be used at least 3 weeks prior to the study (women only), during the infusion period of study drug (men and women), 4-weeks after study drug administration (men and women) and the remaining 11 months in the study follow-up (women). Women must have a negative pregnancy test at screening.
* No greater than mild pericardial effusion < 0.5 cm on echocardiography (roughly corresponds to < 100 mL).
* Have an implantable cardioverter-defibrillator (ICD). The ICD should have been implanted at least 3 months prior to receiving study medication. Patients should undergo interrogation of their ICDs between 1 and 7 days before randomization to drug for the previous thirty (30) days. This interrogation would include surveillance for ventricular arrhythmias as well as assessment of ICD discharge(s) and/or anti-tachycardia pacing.

Exclusion Criteria:

* Has chronic heart failure classified as NYHA Class I or IV.
* Has a history of any malignancy or positive test as specified in the pre-cancer screening.
* Have other conditions which in the opinion of the investigator preclude participation in the study, e.g. serious co-morbidity, known or suspected substance abuse or non-compliance.
* Has a body weight >350lbs.
* Has had any cause hospitalization 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LVEF | 30 days
  Compared to baseline and placebo

SECONDARY OUTCOMES:
Six (6) minute walk test | Day 30, 90, 180, 365
  Compared to baseline and placebo
Quality of Life Questionnaire (Kansas City Cardiomyopathy Questionnaire) | Day 30, 90, 180 and 365
  Compared to baseline and placebo
NYHA class status | Day 30, 90, 180 and 365
  Compared to baseline and placebo
All cause mortality and all cause hospitalization | Days 30, 90, 180 and 365
  Compared to baseline and placebo
Change in LVESV and LVEDV | Day 30
  Compared to baseline and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Barry Greenberg, MD, Study Chair — University of California, San Diego; Uri Elkayam, MD, Principal Investigator — LAC+USC Medical Center
Locations (13):
- United States (13):
  - University of California, San Diego, La Jolla, California
  - Metabolic Clinic and Research Center, Los Angeles, California
  - USC Cardiovascular Division, Los Angeles, California
  - Orange County Research Center, Tustin, California
  - University of Colorado Denver, Denver, Colorado
  - Clearwater Cardiovascular & Interventional Consultants, MD, PA, Clearwater, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - MedPharmics, LLC., Kenner, Louisiana
  - Benchmark Research, Metairie, Louisiana
  - East Texas Cardiology, Houston, Texas
  - The Medical Center of Plano, Plano, Texas
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu Y, Li X, Liu X, Zhou M. Neuregulin-1/ErbB signaling and chronic heart failure. Adv Pharmacol. 2010;59:31-51. doi: 10.1016/S1054-3589(10)59002-1. PMID 20933198
- [Background] Jabbour A, Hayward CS, Keogh AM, Kotlyar E, McCrohon JA, England JF, Amor R, Liu X, Li XY, Zhou MD, Graham RM, Macdonald PS. Parenteral administration of recombinant human neuregulin-1 to patients with stable chronic heart failure produces favourable acute and chronic haemodynamic responses. Eur J Heart Fail. 2011 Jan;13(1):83-92. doi: 10.1093/eurjhf/hfq152. Epub 2010 Sep 1. PMID 20810473
- [Background] Gao R, Zhang J, Cheng L, Wu X, Dong W, Yang X, Li T, Liu X, Xu Y, Li X, Zhou M. A Phase II, randomized, double-blind, multicenter, based on standard therapy, placebo-controlled study of the efficacy and safety of recombinant human neuregulin-1 in patients with chronic heart failure. J Am Coll Cardiol. 2010 May 4;55(18):1907-14. doi: 10.1016/j.jacc.2009.12.044. PMID 20430261
- [Background] Liu X, Gu X, Li Z, Li X, Li H, Chang J, Chen P, Jin J, Xi B, Chen D, Lai D, Graham RM, Zhou M. Neuregulin-1/erbB-activation improves cardiac function and survival in models of ischemic, dilated, and viral cardiomyopathy. J Am Coll Cardiol. 2006 Oct 3;48(7):1438-47. doi: 10.1016/j.jacc.2006.05.057. Epub 2006 Sep 14. PMID 17010808